CLINICAL TRIAL: NCT04950205
Title: The Influence of Postoperative Cognitive Function in Patients With Sevoflurane Postconditioning on Carotid Intima Stripped
Brief Title: Influence of Postoperative Cognitive Function in Patients With Sevoflurane Postconditioning on Carotid Intima Stripped
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2021-0107
Record Dates: First submitted 2021-06-14; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Cognitive Dysfunction; Sevoflurane; Carotid Artery Intima Stripped
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane post conditioning group（S1） (Experimental): propofol：0.05～0.1mg/(kg.min) maintain throughout the whole surgery ,1% sevoflurane plus after open Carotid artery until the end of surgery
  Interventions: Drug: Sevoflurane inhalant product
- The control group（P） (No Intervention): propofol：0.05～0.1mg/(kg.min) maintain throughout the whole surgery without sevoflurane

INTERVENTIONS:
Drug: Sevoflurane inhalant product — propofol plus 1% sevoflurane after open Carotid artery until the end of surgery
  Arms: Sevoflurane post conditioning group（S1）

SUMMARY:
Brief summary: In order to get a better clinical plan for brain protection during perioperative anesthesia for high-risk patients - carotid intima stripped. We observing the hemodynamic changes of sevoflurane post-treatment in carotid intima stripped, the comparison of postoperative cognitive function and postoperative radiographic changes.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists（ASA）：II-III
* Aged between 40 and 80 years
* Patients scheduled for surgery of Carotid stenosis under general anaesthesia

Exclusion Criteria:

* Has a history of mental illness can't cooperate,
* Serious heart block or cardiac decompensation or severe sinus slow (HR < 50 times/min),
* The abnormal nerve monitoring in operation, MMES preoperative score < 20 points,
* Any rescue unexpected occurred during the operation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from the 1 day preoperative to the 1 day postoperative MMSE(Mini-mental State Examination) | the 1st day before the surgery；the 1st day after the surgery
  Screening scale of cognitive function。The highest score is 30 points, 27 to 30 were divided into normal, less than 27 divided into cognitive dysfunction。But is not sensitive in the early identification of dementia, especially in mild cognitive impairment is poorer.
Change from the 1 day preoperative to the 1 day postoperative MoCA(Montreal Cognitive Assessment) | Time Frame: the 1st day before the surgery；the 1st day after the surgery
  Screening scale of cognitive function。The highest score is 30 points，Add 1 score, education the following subjects in less than 12 years。Total score less than 26 divided into cognitive dysfunction。Compared with MMSE, more sensitive to mild dementia。

SECONDARY OUTCOMES:
Heart rate | Ten minutes before induction（T0) ,Intraoperative (Before the carotid artery occlusion（T1）), Intraoperative (before open the Carotid artery（T2)，At the end of the surgery when the surgeon completed sewing skin（T3），the 24 hours after the operation（T4）
  Heart rate per minute
Invasive arterial blood pressure | Ten minutes before induction（T0) ,Intraoperative (Before the carotid artery occlusion（T1）), Intraoperative (before open the Carotid artery（T2)，At the end of the surgery when the surgeon completed sewing skin（T3），the 24 hours after the operation（T4）
  Invasive arterial puncture catheter, continuous arterial pressure monitoring
BIS | Ten minutes before induction（T0) ,Intraoperative (Before the carotid artery occlusion（T1）), Intraoperative (before open the Carotid artery（T2)，At the end of the surgery when the surgeon completed sewing skin（T3），the 24 hours after the operation（T4）
  bispectral index
PETCO2 | Ten minutes before induction（T0) ,Intraoperative (Before the carotid artery occlusion（T1）), Intraoperative (before open the Carotid artery（T2)，At the end of the surgery when the surgeon completed sewing skin（T3），the 24 hours after the operation（T4）
  Partial pressure End-Tidal Carbon Dioxide
Cerebral oxygen saturation | Ten minutes before induction（T0) ,Intraoperative (Before the carotid artery occlusion（T1）), Intraoperative (before open the Carotid artery（T2)，At the end of the surgery when the surgeon completed sewing skin（T3），the 24 hours after the operation（T4）
  Cerebral oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Wang B, Li S, Wang C, Zhu J, Jin Y, Sun D, Lang J. Effect of sevoflurane post-conditioning on postoperative cognitive function in carotid endarterectomy patients: a randomized, double-blind, controlled trial. Front Med (Lausanne). 2025 Dec 8;12:1716370. doi: 10.3389/fmed.2025.1716370. eCollection 2025. PMID 41438154